CLINICAL TRIAL: NCT00955955
Title: TRD - 2: A Double-Blind, Placebo Controlled Study of 6(S)-5-MTHF Among SSRI-Resistant Outpatients With Major Depressive Disorder (MDD)
Brief Title: Study of 6(S)-5-MTHF Among Selective Serotonin Reuptake Inhibitor-Resistant Outpatients With Major Depressive Disorder
Acronym: TRD-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: George I. Papakostas (Other)
Collaborators: Pamlab, L.L.C. (Industry)
Responsible Party: Sponsor-Investigator, George I. Papakostas, Director of Treatment Resistant Depression Studies-DCRP, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006P000604 (2)
Record Dates: First submitted 2009-07-30; First posted 2009-08-10 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Depression
Keywords: Depression; Medical food
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 6(S)-5-MTHF(Deplin) (Experimental): Participants will receive 15 mg/day of Deplin, a medical food, for 8 weeks.
  The SPCD approach, is modified and conducted as follows:
  The phase II dataset of interest is limited to patients treated with placebo during phase I who completed phase I, who did not experience a clinical response according to the HDRS-17 during phase I and entered phase II. Drug is compared to placebo in phase II for this patient subset alone.
  The ITT/LOCF data comparing drug and placebo during phase I is combined with the data comparing drug and placebo according to the SPCD model for phase II (see steps 2 and 3 above), and analyzed using the statistical model as described in Fava et al, 2003
  Interventions: Other: 6(S)-5-MTHF(Deplin)
- Placebo/Deplin (Experimental): Participants will receive placebo for the first 4 weeks, and then 15 mg/day of Deplin (6(S)-5-MTHF) for the next 4 weeks.
  The SPCD approach, is modified and conducted as follows:
  The phase II dataset of interest is limited to patients treated with placebo during phase I who completed phase I, who did not experience a clinical response according to the HDRS-17 during phase I and entered phase II. Drug is compared to placebo in phase II for this patient subset alone.
  The ITT/LOCF data comparing drug and placebo during phase I is combined with the data comparing drug and placebo according to the SPCD model for phase II (see steps 2 and 3 above), and analyzed using the statistical model as described in Fava et al, 2003
  Interventions: Other: 6(S)-5-MTHF(Deplin); Other: Placebo
- Placebo/Placebo (Experimental): Participants will receive placebo for both phases of the study.
  The SPCD approach, is modified and conducted as follows:
  The phase II dataset of interest is limited to patients treated with placebo during phase I who completed phase I, who did not experience a clinical response according to the HDRS-17 during phase I and entered phase II. Drug is compared to placebo in phase II for this patient subset alone.
  The ITT/LOCF data comparing drug and placebo during phase I is combined with the data comparing drug and placebo according to the SPCD model for phase II (see steps 2 and 3 above), and analyzed using the statistical model as described in Fava et al, 2003
  Interventions: Other: Placebo

INTERVENTIONS:
Other: 6(S)-5-MTHF(Deplin) — Deplin is a medical food. Patients will take 15 mg/day of deplin.
  Arms: 6(S)-5-MTHF(Deplin); Placebo/Deplin
Other: Placebo — Inactive substance
  Arms: Placebo/Deplin; Placebo/Placebo

SUMMARY:
The purpose of the study is to test whether oral 6(S)-5-MTHF (Deplin) is safe and effective in relieving depression when it is added to standard kinds of antidepressants called serotonin reuptake inhibitors (SSRIs).

DETAILED DESCRIPTION:
The study consists of two phases, each lasting a total of four weeks (8 weeks total), with visits at the DCRP every 10 days. If the subject is eligible, they will be asked to return two weeks later for a baseline visit, when they will be randomly assigned, like a flip of a coin, to one of three treatment groups: a) drug/drug, b) placebo/drug, c) placebo/placebo (a placebo is a pill that looks like a study drug but contains no active medication). They will have a greater than 50% chance of receiving active medication (Deplin) at some point in the 8 week study.

Neither the subject nor the research staff will know which group the subject is in.

All subjects will be asked to take the study medication in the morning, in addition to their ongoing SSRI treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Meet criteria for current Major Depressive Disorder
* Currently taking an SSRI

Exclusion Criteria:

* Pregnant women
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease
* Prior course of MTHF augmentation, or intolerance to MTHF at any dose
* Substance use disorders active within the last six months, any bipolar disorder (current or past), any psychotic disorder (current or past)
* Have failed more than 2 adequate antidepressant trials during the current Major Depressive Episode

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George I. Papakostas, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - University of California San Diego School of Medicine, San Diego, California
  - Rush University Medical Center, Psychiatric Medicine Associates, LLC, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Cincinnati, College of Medicine, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Shelton RC, Pencina MJ, Barrentine LW, Ruiz JA, Fava M, Zajecka JM, Papakostas GI. Association of obesity and inflammatory marker levels on treatment outcome: results from a double-blind, randomized study of adjunctive L-methylfolate calcium in patients with MDD who are inadequate responders to SSRIs. J Clin Psychiatry. 2015 Dec;76(12):1635-41. doi: 10.4088/JCP.14m09587. PMID 26613389
- [Derived] Papakostas GI, Shelton RC, Zajecka JM, Bottiglieri T, Roffman J, Cassiello C, Stahl SM, Fava M. Effect of adjunctive L-methylfolate 15 mg among inadequate responders to SSRIs in depressed patients who were stratified by biomarker levels and genotype: results from a randomized clinical trial. J Clin Psychiatry. 2014 Aug;75(8):855-63. doi: 10.4088/JCP.13m08947. PMID 24813065
- [Derived] Papakostas GI, Shelton RC, Zajecka JM, Etemad B, Rickels K, Clain A, Baer L, Dalton ED, Sacco GR, Schoenfeld D, Pencina M, Meisner A, Bottiglieri T, Nelson E, Mischoulon D, Alpert JE, Barbee JG, Zisook S, Fava M. L-methylfolate as adjunctive therapy for SSRI-resistant major depression: results of two randomized, double-blind, parallel-sequential trials. Am J Psychiatry. 2012 Dec;169(12):1267-74. doi: 10.1176/appi.ajp.2012.11071114. PMID 23212058

RESULTS

PARTICIPANT FLOW:
Groups:
- Deplin/Deplin: Participants will receive 15 mg/day of Deplin (6(S)-5-MTHF) for 8 weeks.
- Placebo/Deplin: Participants will receive placebo for the first 4 weeks, and then 15 mg/day of Deplin (6(S)-5-MTHF) for the next 4 weeks.
- Placebo/Placebo: Both tablets of study medication will be placebo during both phases of the study.
Period: Overall Study
Arm/Group | Deplin/Deplin | Placebo/Deplin | Placebo/Placebo
Started | 19 | 28 | 28
Completed | 17 | 28 | 28
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deplin/Deplin | Placebo/Deplin | Placebo/Placebo | Total
Number analyzed (Participants) | 19 | 28 | 28 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 28 | 28 | 74
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.58 (14.64) | 50.86 (10.58) | 45.39 (11.60) | 48.49 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 20 | 53
  Male | 5 | 9 | 8 | 22
Region of Enrollment [Number; unit: participants]
  United States | 19 | 28 | 28 | 75

OUTCOME MEASURES:

1. Primary Outcome: The 17-item Hamilton Depression Scale (HAM-D-17)
Description: The HAM-D-17 is a multiple choice questionnaire that clinicians may use to rate the severity of a patient's major depression. Items are scored on a scale of zero to four and higher scores indicate greater impairment. This scale is scored by summing the scores on each item and scores can range from 0-68.
  When assessing changes in HAMD score, negative changes indicate improvement (i.e. the score has decreased) and positive scores indicate a worsening of symptoms (i.e. scores have increased).
Time Frame: Baseline and Day 60
Population: The phase II dataset of interest is limited to patients treated with placebo in phase I, completed phase I, did not experience a clinical response and entered phase II. Drug is compared to placebo in phase II for this subset alone. Some patients received Deplin in both phases of the study, but those patients are not included in these analyses.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Adjunct 6(S)-5-MTHF(Deplin) Phase 1: Participants will receive 15 mg/day of Deplin (6(S)-5-MTHF) for 4 weeks.
- Adjunct Placebo Phase 1: Participants will receive placebo for the first 4 weeks
- Adjunct 6(S)-5-MTHF(Deplin) Phase 2: Participants will receive 15 mg of Deplin (6(S)-5-MTHF) for 4 weeks.
- Adjunct Placebo Phase 2: Patients in this group received placebo in both phases of the study for a total of 8 weeks,
- Pooled Deplin: Patients in this group received Deplin at some point during the study. Results are pooled from phase I and II.
- Pooled Placebo: Patients in this group received placebo at some point during the study. Results are pooled from phase I and II.
Arm/Group | Adjunct 6(S)-5-MTHF(Deplin) Phase 1 | Adjunct Placebo Phase 1 | Adjunct 6(S)-5-MTHF(Deplin) Phase 2 | Adjunct Placebo Phase 2 | Pooled Deplin | Pooled Placebo
Number analyzed (Participants) | 19 | 56 | 18 | 21 | 36 | 75
Scores on a scale | -7.4 (5.2) | -4.4 (5.8) | -3.8 (6.2) | -1.7 (4.7) | -5.58 (5.7) | -3.04 (5.3)
Statistical Analysis 1: Comparison: Pooled Deplin vs Pooled Placebo; Hypothesis 1: There will be a statistically significant difference between the two groups in the degree of improvement, as measured by the change in the 17-item Hamilton Depression Rating Scale (HAM-D-17) score from baseline to endpoint, using the sequential parallel comparison design [51]; with a greater degree of reduction in HAM-D-17 scores in the 6(S)-5-MTHF 15 mg qd group than in the placebo group, with the change on placebo being estimated from Trials 1 and 2; Test type: Superiority or Other; p = .05, SPCD; Sequential Parallel Comparison Design (SPCD); Mean Score Reduction = -5.6, Standard Deviation 5.7 — These results reflect the mean score reduction for the pooled Deplin sample

2. Secondary Outcome: The Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR)
Description: This measure is a 16 item self report questionnaire assessing symptoms of depression. For each item, scores range from 0 to 3 with higher scores indicating greater impairment. To score this measure:
  1. Enter the highest score from questions 1-4 (sleep items): ______
  2. Enter score on item 5 ____
  3. Enter the highest score from questions 6-9 (appetite/weight): ______
  4. Enter score on item 10 ____
  5. Enter score on item 11 ____
  6. Enter score on item 12 ____
  7. Enter score on item 13 ____
  8. Enter score on item 14 ____
  9. Enter the highest score from questions 15-16 (psychomotor items): ______
  Total score range 0-27: ______
  When assessing changes in this measure over time, negative means indicate an improvement (i.e. the scores decreased over time) and positive means indicate worsening in functioning.
Time Frame: Baseline and Day 60
Population: Data presented is mean score reduction for the QIDS. The dataset of interest is limited to patients treated with placebo in phase I, did not experience a clinical response and entered phase II. Drug is compared to placebo in phase II for this subset alone.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Adjunct 6(S)-5-MTHF(Deplin) Phase I: Patients who received Deplin (L-methylfolate) for 4 weeks
- Adjunct Placebo Phase I: Patients who received placebo for 4 weeks.
- Adjunct 6(S)-5-MTHF(Deplin) Phase II: Patients received Deplin for 4 weeks.
- Adjunct Placebo Phase II: Patients received placebo for the second 4 weeks of the study. Patients who received placebo in phase 2 also received it in phase 1.
Arm/Group | Adjunct 6(S)-5-MTHF(Deplin) Phase I | Adjunct Placebo Phase I | Adjunct 6(S)-5-MTHF(Deplin) Phase II | Adjunct Placebo Phase II
Number analyzed (Participants) | 19 | 56 | 18 | 21
Scores on a scale | -8.1 (5.3) | -5.7 (5.6) | -1.3 (4.9) | 0.5 (5.0)

ADVERSE EVENTS:
Time Frame: 60 days
Description: Adverse events data was collected using the SAFTEE measure. Adverse events are reported across both phases of the study. They reflect the number of people who took either medication at any point in the study, not the total number of study participants.
Groups:
- Deplin: Participants will receive 15 mg/day of Deplin (6(S)-5-MTHF).
- Placebo: Adverse events for participants who received placebo during the study.
Arm/Group | Deplin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/54
Other Adverse Events (participants affected / at risk) | 24/42 | 48/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deplin (N=42) | Placebo (N=54)
Gastrointestinal (Gastrointestinal disorders) | 7 (12) | 8 (23)
Sleep (General disorders) | 1 (5) | 3 (12)
Psychological (Psychiatric disorders) | 4 (4) | 9 (12)
Somatic (General disorders) | 6 (12) | 16 (22)
Infectious (Infections and infestations) | 5 (8) | 7 (13)
Miscellaneous (General disorders) | 1 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No